CLINICAL TRIAL: NCT05850598
Title: Effect of Low-frequency rTMS of the Cerebellum on Parkinson's Disease
Brief Title: Effect of rTMS of the Cerebellum on Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Collaborators: Nanjing University (Other)
Responsible Party: Principal Investigator, Pan Yang, Assistant Director Physician, Jiangsu Province Nanjing Brain Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDTMS
Record Dates: First submitted 2023-04-24; First posted 2023-05-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham stimulation targeting the cerebellum (Sham Comparator): Patients will be randomly allocated into this group, and they will receive sham stimulation.
  Interventions: Device: sham rTMS
- real rTMS targeting the cerebellum (Active Comparator): Patients will be randomly allocated into this group, and they will receive real stimulation.
  Interventions: Device: active rTMS

INTERVENTIONS:
Device: sham rTMS — The coil was held while disconnected from the stimulator, and rTMS noise was presented with computer loudspeakers with recorded sound from a real stimulation (20 minutes for each side of the lateral cerebellum everyday for 2 weeks).
  Arms: sham stimulation targeting the cerebellum
Device: active rTMS — Low-frequency (1 Hz) rTMS at with a stimulation intensity of 95% of the motor threshold will be delivered over the bilateral cerebellum for patients with Parkinson's disease (20 minutes for each side of the lateral cerebellum everyday for 2 weeks).
  Arms: real rTMS targeting the cerebellum

SUMMARY:
The goal of this clinical trial is to learn about the efficacy of low-frequency rTMS of the cerebellum in Parkinson's disease.

DETAILED DESCRIPTION:
The main question it aims to answer is: how to improve Parkinson's disease by rTMS.

Participants will be treated with active low-frequency rTMS/sham rTMS over the cerebellum and receive: 1) resting state functional magnetic resonance imaging (fMRI), 2) blood sampling, and 3) Unified Parkinson Disease Rating Scale (UPDRS) before and after the treatment course.

Researchers will compare the data collected from fMRI scan, blood sample analysis, and UPDRS rating between the active rTMS group and sham controls before and after the treatment to see if there are meliorating effects of rTMS on Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Parkinson's disease according to the clinical diagnostic criteria for Parkinson's disease (2015 edition) by the Movement Disorder Society (MDS)
2. Citizens of the People's Republic of China of either sex, aged between 40 and 80 years.
3. Able to give informed consent and follow the research plan.
4. Hoehn-Yahr (H-Y) stage ≤ 3
5. Patients received a Parkinson's stable medication before treatment (assessed via self report), which continued during treatment.

Exclusion Criteria:

1. History or diagnosis of severe psychiatric disorders, such as depression, anxiety disorders, schizophrenia spectrum disorders, and bipolar disorders.
2. Subjects with a clinically defined neurological disorder (assessed via self report) including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, history of stroke, transient ischemic attack within two years, cerebral aneurysm, dementia, multiple sclerosis.
3. Significant cognitive disorders (Mini-Mental State Exam (MMSE)<24 points) or unable to complete the questionnaire independently.
4. Intracranial implants, such as cochlear implants, aneurysms clips, shunts, stimulators, electrodes, cardiac pacemakers and vagus nerve stimulation devices.
5. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold (assess via self report).
6. Showed significant discomfort after receiving the rTMS treatment.
7. Participated in other clinical trials.
8. Inability to read or understand Chinese.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Changes of Unified Parkinson's Disease Rating Scale (UPDRS) (version 3.0) score by rTMS treatment | Baseline, 2 weeks, and 3 months after rTMS treatment
  UPDRS score will be collected from each participants to measure the severity and progression of Parkinson's disease with scores ranging from 0 (minimum) to 199 (maximum). The higher scores mean a worse outcome.
Changes of brain plasticity by rTMS treatment | Baseline, 2 weeks, and 3 months after rTMS treatment
  Resting state fMRI will be scanned from each participants, and brain activity as well as fuctional connectivity will be analyzed.
Changes of circulating serum level of inflammatory cytokines (e.g., Interleukin-1beta (IL-1β), Interleukin-6 (IL-6), and tumor necrosis factor alpha (TNF-α)) by rTMS treatment | Baseline, 2 weeks, and 3 months after rTMS treatment
  Blood samples will be collected from each participants, and serum levels of IL-1β, IL-6, and TNF-α will be measured by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Yang Pan, M. D., Principal Investigator — Jiangsu Province Nanjing Brain Hospital
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No